CLINICAL TRIAL: NCT05699382
Title: Improvement in Mental Health Markers Among Hospital Physicians Through a Mindfulness-training Mobile Application - Randomized Controlled Trial
Brief Title: Improvement Mental Health Among Physicians by a Mindfulness-training Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, yonatan butbul MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0150-20-RMB
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a study group (SG) in which participants practiced mindfulness through the application for 6 weeks (Active Comparator): a study group (SG) in which participants practiced mindfulness through the application for 6 weeks
  Interventions: Other: practiced mindfulness through the application for 6 weeks
- control group (No Intervention): Waiting for the intervention

INTERVENTIONS:
Other: practiced mindfulness through the application for 6 weeks — Physicians working at a tertiary hospital were recruited and randomly divided into two groups, a study group (SG) in which participants practiced mindfulness through the application for 6 weeks
  Arms: a study group (SG) in which participants practiced mindfulness through the application for 6 weeks

SUMMARY:
The aim of our study was to evaluate the effect of a short, smartphone-based mindfulness application on stress, wellbeing and burnout among hospital physicians

DETAILED DESCRIPTION:
Physicians working at a tertiary hospital were recruited and randomly divided into two groups, a study group (SG) in which participants practiced mindfulness through the application for 6 weeks and a control group (CG). Main Measures: All participants filled-out questionnaires assessing stress (Perceived Stress Scale-PSS), mental health (Mental Health Inventory-MHI) and burnout (Maslach Burnout Inventory-MBI) at baseline and 7 weeks later

ELIGIBILITY:
Inclusion Criteria:

* Physicians Working full-time at the Rambam Healthcare Campus.

Exclusion Criteria:

* Physicians that won't be able to participate in at least 50% of the practicing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale-PSS | 7 weeks
  Differences in stress between baseline and 7 weeks later - will be assessed by Perceived Stress Scale-PSS

SECONDARY OUTCOMES:
Mental Health Inventory-MHI | 7 weeks
  Differences in Mental health between baseline and 7 weeks later will be assessed by Mental Health Inventory-MHI
Maslach Burnout Inventory - MBI | 7 weeks
  Differences in Burn out between baseline and 7 weeks later will be assessed by Maslach Burnout Inventory - MBI

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Butbul, Principal Investigator — Rambam
Locations (1):
- Pediatric rheumatology clinic, Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Will be available on request